CLINICAL TRIAL: NCT05811208
Title: Use of Automated Pupillometry for Pain Assessment in ICU Patients with Delirium
Brief Title: Use of Pupillometry for Pain Assessment in ICU Patients with Delirium
Status: Recruiting | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Ivan Cundrle, Clinical Professor, St. Anne's University Hospital Brno, Czech Republic
Other Study IDs: 11V/2023
Record Dates: First submitted 2023-03-30; First posted 2023-04-13 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Delirium; Pain, Postoperative
Keywords: pupillometry; delirium; pain
MeSH Terms: conditions — Delirium; Pain, Postoperative; Pain | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- surgical ICU patients: All surgical patients on the inpatient ward in the Department of Anesthesiology and Intensive Care
  Interventions: Device: automated pupillometry; Diagnostic Test: questionnaire

INTERVENTIONS:
Device: automated pupillometry — Automated pupillometry every 6 hours
Diagnostic Test: questionnaire — CAM ICU questionnaire will be used for delirium screening the incidence of pain will be assessed using 3 valid scales. The Visual Analogue Scale (VAS), the Behavioral Pain Scale (BPS) and the Critical Care Observational Tool (CPOT) will be used.
  questionnaires will be done the same time as pupillometry

SUMMARY:
Pain assessment in intensive care patients is a constant challenge. Approximately 50% to 80% of patients report pain at rest or during medical or nursing interventions (for example endotracheal suctioning, mobilization and rehabilitation, presence and care of invasive inputs, etc.). Obstacles to pain assessment and management are most often due to interference with communication due to impaired consciousness, airway support and connection to artificial pulmonary ventilation, or the effect of administered medication.

Patients in intensive care are prone to delirium. Delirium can compromise patients' ability to verbalise pain for a variety of reasons (e.g. due to impaired attention, memory, thinking and language barriers). Also, pain and inadequate analgesia are risk factors for delirium.

Pupillary reflex changes and their identification by automated pupillometry have yielded positive results regarding nociception assessment in adult and pediatric patients and in perioperative and postoperative care. At the same time, the response of these patients to opioid administration was investigated. The aim was to improve their analgesia.

The aim of this study is to find out whether, there is an association between automated pupillometry and selected objective pain measurement scales in The Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) positive patients after surgery.

DETAILED DESCRIPTION:
Periodically after 6 hours, the incidence of delirium will be assessed using the CAM ICU questionnaire. Subsequently, the incidence of pain will be assessed using 3 valid scales. The Visual Analogue Scale (VAS), the Behavioral Pain Scale (BPS) and the Critical Care Observational Tool (CPOT) will be used. Finally, automated pupillometry will be measured. The measurement values will be entered in the record sheet. Information about the medications administered and the patient's vital signs will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patient after surgery
* possibility to perform CAM - ICU test (patients with Richmond Agitation-Sedation Scale -2 to +2)

Exclusion Criteria:

* eye diseases
* brain injury
* stroke
* epilepsy
* neuromuscular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: surgical patinets admited to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
pupillometry parameters and objective pain scales | up to 4 weeks
  correlation of pupillometry parameters and objective pain scales

CONTACTS AND LOCATIONS:
Overall Officials: Patrik Mica, MSc, Principal Investigator — St. Anne's University Hospital
Locations (1):
- St. Anne's University Hospital in Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alvarez EA, Parada FJ. Association of Pain During the Evaluation of Delirium in Intensive Care Unit Patients. Front Med (Lausanne). 2021 Aug 24;8:722001. doi: 10.3389/fmed.2021.722001. eCollection 2021. No abstract available. PMID 34504855
- [Background] Azevedo-Santos IF, DeSantana JM. Pain measurement techniques: spotlight on mechanically ventilated patients. J Pain Res. 2018 Nov 21;11:2969-2980. doi: 10.2147/JPR.S151169. eCollection 2018. PMID 30538536
- [Background] Fischer T, Hosie A, Luckett T, Agar M, Phillips J. Strategies for Pain Assessment in Adult Patients With Delirium: A Scoping Review. J Pain Symptom Manage. 2019 Sep;58(3):487-502.e11. doi: 10.1016/j.jpainsymman.2019.05.020. Epub 2019 Jun 10. PMID 31195076
- [Background] Rijkenberg S, van der Voort PH. Can the critical-care pain observation tool (CPOT) be used to assess pain in delirious ICU patients? J Thorac Dis. 2016 May;8(5):E285-7. doi: 10.21037/jtd.2016.03.32. No abstract available. PMID 27162683
- [Background] Favre E, Bernini A, Morelli P, Pasquier J, Miroz JP, Abed-Maillard S, Ben-Hamouda N, Oddo M. Neuromonitoring of delirium with quantitative pupillometry in sedated mechanically ventilated critically ill patients. Crit Care. 2020 Feb 24;24(1):66. doi: 10.1186/s13054-020-2796-8. PMID 32093710
- [Background] Tosi F, Gatto A, Capossela L, Ferretti S, Mancino A, Curatola A, Chiaretti A, Pulitano S. Role of the pupillometer in the assessment of pain in the sedation of pediatric patients. Eur Rev Med Pharmacol Sci. 2021 Oct;25(20):6349-6355. doi: 10.26355/eurrev_202110_27008. PMID 34730216
- [Background] Lukaszewicz AC, Dereu D, Gayat E, Payen D. The relevance of pupillometry for evaluation of analgesia before noxious procedures in the intensive care unit. Anesth Analg. 2015 Jun;120(6):1297-300. doi: 10.1213/ANE.0000000000000609. PMID 25993266